CLINICAL TRIAL: NCT00570778
Title: A Randomized, Double-blind, Placebo Controlled, Multicentre Study to Determine the Effect of QVA149 on Lung Function in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy and Safety of QVA149 in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CQVA149A2204
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Results first posted 2013-02-28 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: QVA, Indacaterol, Glycopyrrolate, Concept1, COPD, cross over study, safety and efficacy, trough FEV1
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Glycopyrrolate; indacaterol-glycopyrronium combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- indacaterol/glycopyrrolate 300/50 μg (Experimental): One indacaterol/glycopyrrolate 300/50 μg capsule + 1 placebo capsule inhaled once daily via a single dose dry powder inhaler for 7 days.
  Interventions: Drug: indacaterol/glycopyrrolate
- indacaterol 600 μg (Active Comparator): Two indacaterol 300 μg capsules inhaled once daily via a single dose dry powder inhaler for 7 days.
  Interventions: Drug: indacaterol
- indacaterol 300 μg (Active Comparator): One capsule indacaterol 300 μg + one placebo capsule inhaled once daily via a single dose dry powder inhaler for 7 days.
  Interventions: Drug: indacaterol
- placebo (Placebo Comparator): Two placebo capsules inhaled once daily via a single dose dry powder inhaler for 7 days.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: indacaterol/glycopyrrolate — Inhalation capsule indacaterol/glycopyrrolate 300/50 μg inhaled once daily via a single dose dry powder inhaler for 7 days.
  Other Names: QVA149
  Arms: indacaterol/glycopyrrolate 300/50 μg
Drug: indacaterol — Inhalation capsule indacaterol supplied as 300 μg capsules inhaled once daily via a single dose dry powder inhaler for 7 days.
  Other Names: QAB149
  Arms: indacaterol 300 μg; indacaterol 600 μg
Drug: placebo — Placebo inhalation capsules inhaled once daily via a single dose dry powder inhaler for 7 days.
  Arms: placebo

SUMMARY:
This study will evaluate the safety and efficacy of QVA149 in patients with moderate to severe COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults aged ≥40 years, who have signed an Informed Consent Form prior to initiation of any study-related procedure.
2. Patients with moderate to severe stable Chronic Obstructive Pulmonary Disease (COPD) according to the Global Initiative for Obstructive Lung Disease (GOLD) Guidelines 2006.
3. Patients who have smoking history of at least 10 pack years.
4. Patients with a post-bronchodilator Forced Expiratory Volume in 1 second (FEV1) ≥30% and < 80% of the predicted normal and post-bronchodilator FEV1/Forced Vital Capacity (FVC) <0.70.

Exclusion Criteria:

1. Pregnant or nursing women, or women of child-bearing potential, regardless of whether or not sexually active if they are not using acceptable methods of contraception.
2. Patients requiring long term oxygen therapy (> 15 hours a day) on a daily basis for chronic hypoxemia, or who have been hospitalized or visited an emergency department for a COPD exacerbation or as result of their airways disease in the 6 weeks prior to screening.
3. Patients who have had a respiratory tract infection within 6 weeks prior to screening.
4. Patients with concomitant pulmonary disease, pulmonary tuberculosis (unless confirmed by chest x-ray to be no longer active) or clinically significant bronchiectasis.
5. Patients with any history of asthma indicated by (but not limited to) a blood eosinophil count > 400/mm3.
6. Patients who, in the judgment of the investigator or the responsible Novartis personnel, have a clinically relevant laboratory abnormality or a clinically significant condition.
7. Patients with uncontrolled Type I and Type II diabetes.
8. History of malignancy of any organ system (including lung cancer), treated or untreated, within the past 5 years.
9. Patients who are contraindicated for or who have shown an untoward reaction to inhaled anticholinergic agents.
10. Patients with a history of long QT syndrome or whose QTc interval (Fridericia method) measured at screening is prolonged (>450 ms for males or >470 ms for females).
11. Patients with a history of untoward reactions to sympathomimetic amines, inhaled medication or any component thereof, or any of the study drugs or drugs with similar chemical structures.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (22):
- United States (3):
  - Novartis Investigator Site, St Louis, Missouri
  - Novartis Investigator Site, Charlotte, North Carolina
  - Novartis Investigator site, Raleigh, North Carolina
- Belgium (4):
  - Novartis Investigator Site, Antwerp
  - Novartis Investigator Site, Ghent
  - Novartis Investigator Site, Jambes
  - Novartis Investigator Site, Sankt Vith
- Canada (3):
  - Novartis Investigator Site, Moncton
  - Novartis Investigator Site, Montreal
  - Novartis Investigator site, Toronto
- Germany (6):
  - Novartis Investigator Site, Bad Wörishofen
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Frankfurt
  - Novartis Investigator Site, Mainz
  - Novartis Investigator Site, Rüdersdorf
  - Novartis Investigator Site, Wiesbaden
- Netherlands (6):
  - Novartis Investigator Site, Almelo
  - Novartis Investigator Site, Breda
  - Novartis Investigator site, Eindhoven
  - Novartis investigator site, Heerlen
  - Novartis Investigator Site, Nijmegen
  - Novartis Investigator Site, Veldhoven

REFERENCES:
- [Derived] van Noord JA, Buhl R, Laforce C, Martin C, Jones F, Dolker M, Overend T. QVA149 demonstrates superior bronchodilation compared with indacaterol or placebo in patients with chronic obstructive pulmonary disease. Thorax. 2010 Dec;65(12):1086-91. doi: 10.1136/thx.2010.139113. Epub 2010 Oct 26. PMID 20978028

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was 4 arm crossover study. There was a 7 day washout period between each treatment period. 154 patients were randomized, 153 participants received study drug. 5 patients were excluded from the Modified Intent-to-treat population (MITT). 4 patients for protocol violations and 1 patient was randomized but did not receive study drug.
Groups:
- A: Ind 300 μg- Ind 600 μg- Placebo- Ind/Glyc 300/50 μg: Treatment Period 1: One indacaterol (Ind) 300 μg capsule and one placebo capsule inhaled once daily via a single dose dry powder inhaler (SDDPI) for 7 days.
  Treatment Period 2: Two indacaterol 300 μg capsules inhaled once daily via a SDDPI for 7 days.
  Treatment Period 3: Two placebo capsules inhaled once daily via a SDDPI for 7 days.
  Treatment Period 4: One indacaterol/glycopyrrolate (Ind/Glyc) 300/50 μg and one placebo capsule inhaled once daily via a SDDPI for 7 days.
- B: Ind 600 μg- Placebo- Ind/Glyc 300/50 μg- Ind 300 μg: Treatment Period 1: Two indacaterol 300 μg capsules inhaled once daily via a SDDPI for 7 days.
  Treatment Period 2: Two placebo capsules inhaled once daily via a SDDPI for 7 days.
  Treatment Period 3: One indacaterol/glycopyrrolate (Ind/Glyc) 300/50 μg and one placebo capsule inhaled once daily via a SDDPI for 7 days.
  Treatment Period 4: One indacaterol (Ind) 300 μg capsule and one placebo capsule inhaled once daily via a SDDPI for 7 days.
- C: Ind/Glyc 300/50 μg- Ind 300 μg- Ind 600 μg- Placebo: Treatment Period 1: One indacaterol/glycopyrrolate (Ind/Glyc) 300/50 μg and one placebo capsule inhaled once daily via a SDDPI for 7 days.
  Treatment Period 2: One indacaterol (Ind) 300 μg capsule and one placebo capsule inhaled once daily via a SDDPI for 7 days.
  Treatment Period 3: Two indacaterol 300 μg capsules inhaled once daily via a SDDPI for 7 days.
  Treatment Period 4: Two placebo capsules inhaled once daily via a SDDPI for 7 days.
- D: Placebo- Ind/Glyc 300/50 μg- Ind 300 μg- Ind 600 μg: Treatment Period 1: Two placebo capsules inhaled once daily via a SDDPI for 7 days.
  Treatment Period 2: One indacaterol/glycopyrrolate (Ind/Glyc) 300/50 μg and one placebo capsule inhaled once daily via a SDDPI for 7 days.
  Treatment Period 3: One indacaterol (Ind) 300 μg capsule and one placebo capsule inhaled once daily via a SDDPI for 7 days.
  Treatment Period 4: Two indacaterol 300 μg capsules inhaled once daily via a SDDPI for 7 days.
Period: Overall Study
Arm/Group | A: Ind 300 μg- Ind 600 μg- Placebo- Ind/Glyc 300/50 μg | B: Ind 600 μg- Placebo- Ind/Glyc 300/50 μg- Ind 300 μg | C: Ind/Glyc 300/50 μg- Ind 300 μg- Ind 600 μg- Placebo | D: Placebo- Ind/Glyc 300/50 μg- Ind 300 μg- Ind 600 μg
Started | 41 | 38 | 37 | 38
Safety Population: Received Study Drug | 41 (Safety Population included all participants who received at least 1 dose of any study drug.) | 38 | 36 | 38
Modified Intent-to-treat Population | 40 | 37 | 35 | 37
Completed | 37 | 34 | 30 | 34
Not Completed | 4 | 4 | 7 | 4
Not completed — Protocol deviation | 2 | 1 | 2 | 2
Not completed — Adverse Event | 0 | 1 | 4 | 1
Not completed — Subject withdrew consent | 0 | 1 | 0 | 1
Not completed — Abnormal test procedure | 1 | 0 | 0 | 0
Not completed — Unsatisfactory therapeutic effect | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Subject no longer requires study drug | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Population: Participants were randomized and received the following 4 treatments: 1-Two placebo capsules inhaled once daily via a SDDPI for 7 days, 2-One indacaterol/glycopyrrolate (Ind/Glyc) 300/50 μg and one placebo capsule inhaled once daily via a SDDPI for 7 days, 3-One Indacaterol (Ind) 300 μg capsule and one placebo capsule inhaled once daily via a SDDPI for 7 days and 4-Two Indacaterol 300 μg capsules inhaled once daily via a SDDPI for 7 days. There was a 7 day washout period between the four treatment periods.
Arm/Group | Overall Population
Number analyzed (Participants) | 153
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline characteristics are based on the Safety Population that consists of all participants who received study drug.
  years | 61.7 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 94

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) at Day 7
Description: Spirometry testing was performed in accordance with American Thoracic Society standards. Trough FEV1 was defined as the average of the 23 hour 15 minute and 23 hour 45 minute measurements post dosing. Baseline FEV1 is the mean of the 45 minute and 15 minute pre-dose FEV1 values at day 1 of each period. Least square means are based on the Analysis of Covariance Trough FEV1 at day 7 = sequence effect + patient(sequence) + period effect + treatment effect + (period) baseline FEV1 + error.
Time Frame: Baseline, Day 7
Population: Participants from the Modified Intent-to-treat population (includes all participants who received study drug) with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol/Glycopyrrolate 300/50 μg | Indacaterol 300 μg | Indacaterol 600 μg | Placebo
Number analyzed (Participants) | 140 | 138 | 140 | 136
Liters | 1.512 (0.0143) | 1.389 (0.0144) | 1.395 (0.0143) | 1.286 (0.0145)

2. Secondary Outcome: Standardized Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve (AUC) 5 Minutes-12 Hours at Day 7
Description: Spirometry testing was performed in accordance with American Thoracic Society standards. FEV1 was assessed at 5, 15, 30 minutes, 1, 2, 3, 4, 5, 6, 8, 10 and 12 hours post dose on Day 7. Standardized (with respect to time) AUC (5 minutes-12 hours) for FEV1 on day 7 was calculated using the trapezoidal rule. Least square means are based on the Analysis of Covariance: FEV1 AUC = sequence effect + patient (sequence) + period + treatment + baseline FEV1 (period) + error.
Time Frame: Day 7
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol/Glycopyrrolate 300/50 μg | Indacaterol 300 μg | Indacaterol 600 μg | Placebo
Number analyzed (Participants) | 142 | 140 | 142 | 140
Liters | 1.610 (0.0180) | 1.473 (0.0181) | 1.457 (0.0180) | 1.317 (0.0185)

3. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Discontinuations Due to Adverse Events
Description: Additional information about adverse events can be found in the Adverse Event Section.
Time Frame: 47 days
Population: Safety population includes all participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Indacaterol/Glycopyrrolate 300/50 μg | Indacaterol 300 μg | Indacaterol 600 μg | Placebo
Number analyzed (Participants) | 142 | 141 | 141 | 143
Participants
  Serious Adverse Events | 2 | 0 | 0 | 0
  Adverse Events | 39 | 31 | 37 | 31
  Discontinuations Due to Adverse Events | 3 | 0 | 2 | 0

ADVERSE EVENTS:
Description: The number of patients in the safety population for the QAB 600 μg treatment is (N=141) compared to the safety population (N=142). One patient was mistakenly dosed with QAB149 600 μg in 2 out of 4 periods. For AEs, this patient was counted once, not twice, therefore the difference in one patient.
Groups:
- Indacaterol/Glycopyrrolate 300/50 μg: One indacaterol/glycopyrrolate 300 μg /50 μg capsule + 1 placebo capsule inhaled once daily via a single dose dry powder inhaler for 7 days.
Arm/Group | Indacaterol/Glycopyrrolate 300/50 μg | Indacaterol 300 μg | Indacaterol 600 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/142 | 0/141 | 0/141 | 0/143
Other Adverse Events (participants affected / at risk) | 12/142 | 14/141 | 15/141 | 15/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol/Glycopyrrolate 300/50 μg (N=142) | Indacaterol 300 μg (N=141) | Indacaterol 600 μg (N=141) | Placebo (N=143)
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol/Glycopyrrolate 300/50 μg (N=142) | Indacaterol 300 μg (N=141) | Indacaterol 600 μg (N=141) | Placebo (N=143)
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 2 | 2
Nasopharyngitis (Infections and infestations) | 1 | 6 | 2 | 5
Headache (Nervous system disorders) | 7 | 2 | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.